CLINICAL TRIAL: NCT00737984
Title: Improving the Pregnancy Rate With Endometrial Sampling Before Intrauterine Insemination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because very low number of patients were enrolled
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Mohammed Agdi, Consultant Reproductive Endocrinology and Infertility, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDR-08-004
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2009-10

CONDITIONS: Infertility; Clinical Pregnancy Rate
Keywords: Infertility; Clinical pregnancy rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Group 1 patients will receive standard superovulation-IUI treatment without endometrial sampling
- 2 (Active Comparator): Group 2 patients will receive standard superovulation-IUI treatment with endometrial sampling performed in the preceding cycle. It will be done in the follicular phase not later than day 10 of the cycle
  Interventions: Procedure: Endometrial sampling

INTERVENTIONS:
Procedure: Endometrial sampling — Endometrial sampling performed in the preceding cycle. It will be done in the follicular phase not later than day 10 of the cycle
  Other Names: Intrauterine insemination; Clinical pregnancy rate
  Arms: 2

SUMMARY:
Endometrial sampling improves the pregnancy rates in superovulation-IUI cycles

DETAILED DESCRIPTION:
Endometrial sampling is performed using the standard technique in the outpatient department. Similarly, superovulation with gonadotrophins will be performed according to our standard practice.Endometrial sampling will be done in the follicular phase not later than day 10 of the cycle. Endometrial sampling will be performed using Pipelle sampling catheter. The Pipelle is inserted gently through the cervical canal into the uterine cavity and advanced slowly till just resistance felt by the operator. Then, the piston is withdrawn to create negative suction and gentle movement of Pipelle up and down in the uterine cavity is performed while it is against the uterine wall. The Pipelle catheter is withdrawn gently and any obtained specimen will be sent for histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

1. All women undergoing superovulation with gonadotrophins and intrauterine insemination.
2. All women with cervical factor, mild male factor and/or unexplained infertility.
3. At least one patent Fallopian tube.

Exclusion Criteria:

1. Bilateral tubal disease
2. Severe male factor infertility
3. Intrauterine pathology (submucosal fibroid, endometrial polyp, adhesions)
4. Women with positive cervical culture and/or acute vaginal infection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The rate of clinical pregnancy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Togas Tulandi, MD, MHCM, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Background] Raziel A, Schachter M, Strassburger D, Bern O, Ron-El R, Friedler S. Favorable influence of local injury to the endometrium in intracytoplasmic sperm injection patients with high-order implantation failure. Fertil Steril. 2007 Jan;87(1):198-201. doi: 10.1016/j.fertnstert.2006.05.062. PMID 17197286
- [Result] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877